CLINICAL TRIAL: NCT05172518
Title: Utidelone Plus Capecitabine Versus Taxane Plus Capecitabine in HER2-negative Locally Advanced or Metastatic Breast Cancer : A Phase III, Open-label, Randomized Controlled Trial
Brief Title: Utidelone Plus Capecitabine Versus Taxane Plus Capecitabine in HER2-negative Locally Advanced or Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chengdu Biostar Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-2021-UCAN
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Breast Neoplasms; Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — taxane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Active Comparator): Taxane plus Intermittent Capecitabine
  Interventions: Drug: Taxane plus Intermittent Capecitabine
- Arm B (Experimental): Utidelone plus Intermittent Capecitabine
  Interventions: Drug: Utidelone plus Intermittent Capecitabine
- Arm C (Active Comparator): Taxane plus Metronomic Capecitabine
  Interventions: Drug: Taxane plus Metronomic Capecitabine
- Arm D (Experimental): Utidelone plus Metronomic Capecitabine
  Interventions: Drug: Utidelone plus Metronomic Capecitabine

INTERVENTIONS:
Drug: Taxane plus Intermittent Capecitabine — Eligible patients will receive treatment with taxane (paclitaxel, nab-paclitaxel or docetaxel , the dosage reference to related prescribing information or clinical practice by investigators) plus capecitabine (1000 mg/ m2 twice daily D1-14 Q3W) for 6 ~8 cycles(for the the patients with SD, PR or CR after 6~8 cycles treatment could choose to receive continuous combination therapy or capecitabine maintenance mono therapy ), or be treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm A
Drug: Utidelone plus Intermittent Capecitabine — Eligible patients will receive treatment with utidelone (30 mg/ m2 /day D1-5 Q3W) plus capecitabine (1000 mg/ m2 twice daily D1-14 Q3W) for 6 ~8 cycles(for the the patients with SD, PR or CR after 6~8 cycles treatment could choose to receive continuous combination therapy or capecitabine maintenance mono therapy), or be treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm B
Drug: Taxane plus Metronomic Capecitabine — Eligible patients will receive treatment with taxane (paclitaxel, nab-paclitaxel or docetaxel , the dosage reference to related prescribing information or clinical practice by investigators) plus capecitabine ( 500 mg three times daily on days 1-21 Q3W) for 6 ~8 cycles(For the the patients with SD, PR or CR after 6~8 cycles treatment could choose to receive continuous combination therapy or capecitabine maintenance mono therapy), or be treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm C
Drug: Utidelone plus Metronomic Capecitabine — Eligible patients will receive treatment with utidelone (30 mg/ m2 /day D1-5 Q3W) plus capecitabine (500 mg three times daily on days 1-21 Q3W) for 6 ~8 cycles(for the the patients with SD, PR or CR after 6~8 cycles treatment could choose to receive continuous combination therapy or capecitabine maintenance mono therapy ), or be treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm D

SUMMARY:
It is a phase III trial to explore the efficacy and safety of utidelone plus capecitabine versus taxane plus capecitabine in HER2-negative locally advanced or metastatic breast cancer and the differences of metronomic capecitabine and intermittent capecitabine in combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Women aged ≥ 18 years;
* Patients with locally advanced or metastatic, histologically or cytologically documented breast cancer;
* The primary tumor and metastases (if aspirated) are both HER2-negative;
* Eastern Cooperative Oncology Group (ECOG) score [0-2] points;
* Measurable disease according to RECIST version 1.1;
* Previous chemotherapy with taxane for early breast cancer (eBC; neoadjuvant or adjuvant setting) is permitted if completed ≥12 months before randomisation;
* No more than one prior chemotherapy regimen for inoperable locally advanced or metastatic HER2-negative breast cancer;
* Hormone receptor positive patients are allowed no more than two lines of prior endocrine therapy for metastatic disease (including CDK4/6 inhibitors, chidamide and PI3K inhibitors, etc.);
* Patients must have recovered to ≤ Grade 1 (CTCAE v5.0) from all toxicities related to prior antineoplastic therapy. However, patients with any grade of alopecia are allowed ;
* Patients with asymptomatic CNS metastases may be enrolled, if:

  1. Intracranial lesions are evaluable and eligible for systemic therapy only in the absence of extracranial evaluable lesions, or
  2. Patients with stable intracranial lesions after local treatment while there are extracranial evaluable lesions ;
* Adequate hematological, hepatic and renal function;
* Women of child bearing potential must agree to use a contraceptive method during the treatment period and for at least 90 days after the last dose of experiment treatment;
* Life expectancy of at least 12 weeks;
* Patients must be able to participate and comply with treatment and follow-up.

Exclusion Criteria:

* HER-2 positive (IHC + + +, or FISH positive);
* Other malignancies (including primary brain or leptomeninges-related tumors) within the past 5 years, except cured cutaneous basal cell carcinoma and cervical carcinoma in situ;
* Patients who have received anti-tumor therapy within 4 weeks prior to the start of study treatment, including chemotherapy, radical radiotherapy, hormone therapy, biological therapy, immunotherapy or anti-tumor Chinese medicine therapy;
* Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks before the first dose of treatment, or anticipating for a major surgical procedure during the study;
* Symptomatic peripheral neuropathy or CTCAE 5.0 grade ≥ 2;
* Experienced grade 3 or above nervous system-related adverse events after treatment with anti-microtubule drugs;
* Received taxane and/or capecitabine-containing adjuvant/neoadjuvant chemotherapy within 1 year prior to the first study treatment;
* Received prior first-line chemotherapy containing a taxane or capecitabine;
* Symptomatic central nervous system metastases;
* Inability to take or absorb oral medications;
* Pregnant or lactating women;
* Known or suspected hypersensitivity to any of the study drugs or excipients;
* Any other non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that precludes study treatment implementation or follow-up ；
* Any other condition that the investigator considers inappropriate to participate in this trial .
* Use of corticosteroids is prohibited.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 60 months
  Time from randomization to progression or death (whichever occurred first).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 60 months
  The proportion of patients with a best response of CR or PR, according to RECIST 1.1 criteria.
Time to response (TTR) | up to 60 months
  the time from randomization to the first documentation of disease response (CR or PR).
Duration of response (DOR) | up to 60 months
  the time from the first evaluation that criteria for CR or PR are met until PD or death is observed, whichever occurs first, calculated only for patients whose best response is evaluated as CR or PR.
Overall survival (OS) | up to 60 months
  Time from randomization to death Time from randomization to death Time from randomization to death Time from randomization to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Shusen Wang, Guangzhou, Guangdong, China